CLINICAL TRIAL: NCT04646603
Title: A Phase IIa, Adaptive, Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study in Hospitalized Patients Infected With Severe and Critical SARS-CoV-2 to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of MRG-001
Brief Title: MRG-001 as an Immunoregulatory and Regenerative Therapy for COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedRegen LLC (Industry)
Collaborators: ICON plc (Industry); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRG2020
Record Dates: First submitted 2020-11-24; First posted 2020-11-30 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; ARDS, Human; Stem Cells; Regeneration
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Double-Blind Randomized Placebo-Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRG-001 (Experimental): Multiple SC dose of 0.0066 mL/kg MRG-001 (n=20) will be administered every other day for the duration of 13 days totaling 7 injections.
  Interventions: Drug: MRG-001
- Placebo (Placebo Comparator): Single SC dose of 0.0066 mL/kg Sterile Injectable Saline (n=20) will be administered every other day for the duration of 13 days totaling 7 injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRG-001 — Subjects will receive subcutaneous MRG-001 injections.
  Arms: MRG-001
Drug: Placebo — Subjects will receive subcutaneous placebo injections.
  Arms: Placebo

SUMMARY:
This study consists of two parts.

Part A (Phase I):

A Phase I Double-blind Randomized Placebo-controlled Study in Healthy Subjects to Assess the Safety, Pharmacokinetics, Pharmacodynamics of MRG-001

Part B (Phase 2):

A Phase IIa, Adaptive, Double-Blind, Randomized, Placebo-controlled, Multi-center Study in Hospitalized Patients Infected with Severe and Critical SARS-CoV-2 to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of MRG-001

DETAILED DESCRIPTION:
MRG-001 is a fixed-dose combination (FDC) drug, administered as a single subcutaneous (SC) injection. Preclinical studies have demonstrated a synergistic effect of these 2 APIs in mobilizing and recruiting stem cells/immunoregulatory cells and promoting tissue regeneration in a wide variety of studies.

MRG-001 is likely to target multiple aspects of the COVID-19. MRG-001 exhibits immunoregulatory and regenerative properties in preclinical studies with a wide variety of diseases. Repairing damaged tissues in the lung and other organs, restoring the anti-virus immune system and modulating the inflammation are obvious therapeutic targets for COVID-19.

Part A has been completed in May 01, 2021.

Part B has been initiated in January 2022.

ELIGIBILITY:
Inclusion Criteria

1. Subject voluntarily agrees to participate in this study and is able to provide written informed consent or has a legal representative who can provide informed consent.
2. Males and females over 18 years of age, inclusive, at the time of signing the ICF.
3. Hospitalized, with COVID-19 symptoms of respiratory illness caused by SARS-CoV-2 infection (defined as Scale 5 - 7 on the WHO 8-point ordinal scale for clinical improvement.
4. Laboratory-confirmation SARS-CoV-2 by real time polymerase chain reaction in the respiratory tract (NP swab, oropharyngeal swab, tracheal aspirate, BAL) </=14 days prior to randomization.
5. Radiologic findings compatible with diagnosis of SARS-CoV-2 pulmonary infection.
6. Women of childbearing potential must be willing and able to use at least one highly effective contraceptive method for a period from the screening visit until the end of study visit.
7. Men must be willing to use a double-barrier contraception from enrollment until at 5 months after the last dose of study drug, if not abstinent.

Exclusion Criteria

1. Participation in any other clinical trial of an experimental treatment for COVID-19 (remdesivir use is permitted).

2. Significant pre-existing organ dysfunction prior to randomization

1. Lung: Receiving supplemental home oxygen therapy at baseline for pre-existing medical condition (other than COVID-19), as documented in medical record
2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record. clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction (past 3 months), heart and coronary vessel surgery (past 3 months), significant valvular heart disease, uncontrolled arterial hypertension with systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg.
3. Renal: End-stage renal disease requiring renal replacement therapy or eGFR <30 mL/min
4. Liver: Severe chronic liver disease defined as Child-Pugh Class C
5. Hematologic: Baseline platelet count <50,000/mm3

   2. Concurrent treatment or prior use of drugs with actual or possible direct acting immunomodulatory activity against ARDS in COVID-19 is prohibited including JAK1/JAK2 inhibitor ruxolitinib, baricitinib and tofacitinib. However, IL-6 inhibitors such as tocilizumab, sarilumab are allowed if given >72 hours prior to first study dose. Corticosteroids are permitted throughout the study.

   3. History of splenectomy or splenomegaly (spleen weighing >750 g).

   4. Body mass index of >45 kg/m2 at screening

   5. Underlying malignancy, or other condition, with estimated life expectancy of less than two months

   6. Known family history of long QT syndrome (Torsades de Pointes) or currently taking medication that prolongs QT interval.

   7. Currently taking immunomodulating biologics (e.g., interferons, interleukin).

   8. Extracorporeal membrane oxygenation (ECMO).

   9. Use of two or more vasopressors.

   10. Female subjects who are pregnant or breastfeeding or planning to breastfeed at any time through 90 days after last dose of IP.

   11. Received a live-attenuated vaccine within 30 days prior to enrollment.

   12. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, human immunodeficiency virus (HIV) antibody or Active tuberculosis or a history of inadequately treated tuberculosis.

   13. Ongoing immunosuppression: solid organ transplant recipients.

   14. Has used an investigational drug within 30 days prior to Screening.

   15. History of hypersensitivity to MRG-001 (plerixafor [AMD3100, 24 mg/mL]) and tacrolimus [FK506, 0.5 mg/mL]) or any of the excipients or to medicinal products with similar chemical structures.

   16. Current treatment with an anti-viral medication for COVID-19 (e.g. hydroxychloroquine, lopinavir/ritonavir), other than remdesivir.

   17. Unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.

   18. Unlikely to comply with the protocol requirements, instructions and study related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.

   19. Previously been enrolled in this clinical study.

   20. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).

   21. Any condition that in the opinion of the treating physician will increase the risk for the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 60 days
  To evaluate the safety (SAE's) of MRG-001 in Severe and Critical SARS-CoV-2 patients.

SECONDARY OUTCOMES:
Change in percentages from baseline in circulating white blood cell subpopulations | 15 days
Change in Plerixafor concentration (ng/ml) from baseline in blood | 15 days
Change in Tacrolimus concentration (ng/ml) from baseline in blood | 15 days
Change from baseline in ALT, AST, INR, Albumin, Bilirubin, LDH, BUN, eGFR | 15 days
Change in percentages from baseline in circulating stem cells and immune cells | 15 days
All-cause mortality assessed at 14, 28 and 60 days following randomization. | 60 days
Time to clinical improvement from randomization by at least 2 points on the 8-point ordinal scale of WHO clinical improvement scale assessed up to 14 and 60 days (1=Asymptomatic, no limitations of activities; 8=death). | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Russell N Wesson, M.B.Ch.B, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be given a unique unidentifiable study ID number and all data will be recorded according to unidentifiable number to protect patients personal health information.

REFERENCES:
- [Derived] Ahmadi AR, Atiee G, Chapman B, Reynolds L, Sun J, Cameron AM, Wesson RN, Burdick JF, Sun Z. A phase I, first-in-human study to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of MRG-001 in healthy subjects. Cell Rep Med. 2023 Sep 19;4(9):101169. doi: 10.1016/j.xcrm.2023.101169. Epub 2023 Aug 25. PMID 37633275